CLINICAL TRIAL: NCT01913249
Title: Effect of Short Term Versus Long Term Treatment With Seton Prior to LIFT Surgery for Complex Anal Fistula, a Randomized Controlled Trial.
Brief Title: Effect of Short Term Versus Long Term Treatment With Seton Prior to LIFT Surgery for Complex Anal Fistula
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to get MRI of patients within reasonable time on a local hospital.
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/581(REK)
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2013-09

CONDITIONS: Anorectal Fistula
Keywords: Anorectal fistula; LIFT; Seton
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Seton through fistula 6 months prior to LIFT
  Interventions: Procedure: LIFT
- Control (Active Comparator): Seton through fistula 3 weeks prior to LIFT surgery
  Interventions: Procedure: LIFT

INTERVENTIONS:
Procedure: LIFT — Ligation of intersphincteric fistula tract

SUMMARY:
The aim of this study is to compare short term (3 week) with long term (6 months) treatment with seton prior to LIFT surgery. The main end-points are recurrence rates and complication rates after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years
* Complex anal fistula defined as

  * anterior fistulas in women
  * branched fistulas
  * fistulas in patients with anal incontinence
  * fistulas traversing more than 30% of the anal sphincter and therefore unsuitable for simple division.

Exclusion Criteria:

* Crohn's disease in the rectum
* Previous LIFT surgery on same side
* Patient already treated with seton > 3 weeks
* Not able or willing to sign informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 1 year
  Recurrence or non-healing of anal fistula one year after LIFT surgery
Complication | 1 year
  Main complication being anal incontinence measured by St.Marks score, but all major and minor complications are registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Sykehuset Innlandet, Hamar, Norway